CLINICAL TRIAL: NCT07119671
Title: Peer-Aid and Hope Box: A Feasibility Study of a Combined Intervention for Suicidal Patients Hospitalized in a Psychiatric Crisis Unit
Brief Title: Peer-aid and Hope Box
Acronym: HOPAIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A00082-47
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Suicide Prevention
Keywords: Suicide prevention; Hope box; Pair aid
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Mixed bi-centric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOPAIR Intervention: Meeting between Peer helper and Concerned Individual in Psychiatric Crisis Unit (Other): This intervention begins with an initial discussion focused on the individual's lived experience, followed by an explanation of the Hope Box's principle, utility, and use. After each intervention, the peer supporter will complete a satisfaction self-questionnaire to provide feedback.
  Interventions: Other: HOPAIR Intervention: Meeting between Peer Helper and Concerned Individual in Psychiatric Crisis Unit

INTERVENTIONS:
Other: HOPAIR Intervention: Meeting between Peer Helper and Concerned Individual in Psychiatric Crisis Unit — This intervention begins with an initial discussion focused on the individual's lived experience, followed by an explanation of the Hope Box's principle, utility, and use. After each intervention, the peer supporter will complete a satisfaction self-questionnaire to provide feedback.

SUMMARY:
Since 2014, suicide prevention has been a national priority and is one of the 3 priority areas of the mental health plan's roadmap .

Hospitalization offers a crucial opportunity for life-preserving intervention . Brief health interventions and contacts are reputed to be easy to implement, effective and inexpensive .

The Hope Box is a practical emotional management tool that aims to encourage the expression of reasons for living by materializing them in a customizable box, filled with objects, photos, writings and memories in order to find comfort and hope .

Peer support use their experiential knowledge of disorders and recovery to accompany people and help humanize care . They can play a decisive role in suicide prevention .

In contrast to an approach focusing only on risk factors, peer support and the Hope Box are both focus on protective factors, the strengths of the people concerned and hope.

The primary objective of this study is to evaluate the feasibility of the HOPAIR intervention (peer-support and Hope Box, completed by a reminder postcard) with suicidal people hospitalized in psychiatric crisis units. Its secondary objective is to assess the potential effectiveness on intensity of hopelessness, sense of self-efficacy, reasons for living, perceived social support and suicidal recurrence at 3 months.

This is a mixed-methods study involving 40 patients and 2 peer support in two crisis hospitalization units.

DETAILED DESCRIPTION:
Around 703,000 people die by suicide each year worldwide, with suicide prevention being a national priority in France since 2014. The period after a patient is discharged from the hospital is a particularly high-risk time for suicide, especially for those with a history of suicide attempts.

This study proposes a new intervention called HOPAIR, which combines three key components:

* Peer support: A professional peer-helper, who has personal experience with mental health challenges, meets with the patient to share their recovery story and foster a sense of hope and connection.
* The Hope Box: A personalized box that patients fill with objects, photos, and memories to engage their five senses and serve as a tool for emotional management, comfort, and distraction during times of distress.
* A reminder postcard: Sent one month after the initial intervention to reinforce the key concepts of the Hope Box and maintain motivation.

The primary objective of the HOPAIR study is to evaluate the feasibility of this combined intervention for suicidal patients hospitalized in a psychiatric crisis unit. The study also aims to assess the potential effectiveness of HOPAIR on several factors after three months, including:

* Feelings of hopelessness and self-efficacy
* Reasons for living
* Perceived social support
* The presence of suicidal thoughts and repeat suicide attempts The study is a mixed-methods, bi-centric research project that will recruit patients 24-48 hours after admission. The intervention will take place within two to four days of admission, followed by the postcard mailing one month later, and a final evaluation at three months. This evaluation will include re-administering scales to measure the study's objectives and conducting qualitative interviews with a subset of participants to assess their satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* Major ;
* Hospitalized in a psychiatric crisis unit;
* Having attempted suicide in the month preceding hospitalisation;
* Able to give free and informed consent;
* Having given consent;
* French-speaking person with at least B1 level (reading and writing);
* With access to the technical resources required for the study;
* With a postal address.

Exclusion Criteria:

* Presenting a relational modality incompatible with the proposed intervention (agitation, acute delirium, major cognitive disorders or psychic disorganisation, etc.);
* Included in another research protocol related to suicide prevention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility Evaluation of the Combined HOPAIR Intervention (Peer Support, Hope Box, and Postcard Reminder) for Suicidal Inpatients in Psychiatric Crisis Units at 3-Month Post-Intervention. | 37 months
  It will be assessed by :
  * Achievement of the target of recruiting two peer support (yes/no).
  * Completion of training by the two peer support (yes/no).
  * Recruitment capacity of 40 patients, 20 in each center;
  * Collection and description of the characteristics of the resulting sample at the time of inclusion by the IPA within 24 hours of arrival in the department;
  * The acceptability of the intervention and the use of the Hope Box through feedback from the people concerned by means of a semi-directive telephone interview at 3 months by the IPA;
  * Feedback from peer support after each intervention, using self-questionnaires;

SECONDARY OUTCOMES:
Effectiveness of the HOPAIR intervention on indicators of well-being at 3 months post-intervention. | 37 months
  The potential effectiveness of the HOPAIR system will be assessed by comparing the differences in scores and responses to questions at inclusion, during a face-to-face interview and at 3 months after the HOPAIR intervention during a telephone interview by the IPA using the following scales and questions.
Effectiveness of the HOPAIR intervention on indicators of suicidality at 3 months post-intervention. | 37 months
  The potential effectiveness of the HOPAIR system will be assessed by comparing the differences in scores and responses to questions at inclusion, during a face-to-face interview and at 3 months after the HOPAIR intervention during a telephone interview by the IPA using the following scales and questions

CONTACTS AND LOCATIONS:
Overall Officials: Tamara VERNET, IPA, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: No